CLINICAL TRIAL: NCT05610839
Title: A Randomized Controlled Trial of a Fully-automated Self-help AEBT Website for Adults With Trichotillomania
Brief Title: A RCT of a Fully-automated Self-help AEBT Website
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13026
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: AEBT Website With Check-ins; AEBT Website Without Check-ins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AEBT website with check-ins (Experimental): Participants will complete the 8-module intervention of Acceptance-enhanced behavior therapy (AEBT) and will receive weekly check-ins. Acceptance-enhanced behavior therapy is a manualized treatment approach created by Woods and Twohig 2008 that provides both Acceptance and Commitment Therapy and Habit Reversal Therapy.
  Interventions: Behavioral: Acceptance-Enhanced Behavior Therapy
- AEBT website without check-ins (Active Comparator): Participants will complete the 8-module intervention of Acceptance-enhanced behavior therapy (AEBT) but will not receive weekly check-ins. Acceptance-enhanced behavior therapy is a manualized treatment approach created by Woods and Twohig 2008 that provides both Acceptance and Commitment Therapy and Habit Reversal Therapy.
  Interventions: Behavioral: Acceptance-Enhanced Behavior Therapy

INTERVENTIONS:
Behavioral: Acceptance-Enhanced Behavior Therapy — 8-module intervention delivering acceptance-enhanced behavior therapy through a fully automated website. This intervention was adapted from the Acceptance-enhanced behavior therapy workbook (Woods & Twohig, 2008).

SUMMARY:
Trichotillomania (TTM) is characterized by hair pulling that is repetitive in nature leading to notable hair loss, causing clinically significant distress and resulting in impairments across social and functional domains (APA, 2013). Trichotillomania causes significant social impairment including affecting close relationships, pursuing occupational changes or advancement, or interfering with schooling (Grant et al., 2017; Woods, Flessner, Franklin, Wetterneck, et al., 2006). The core of the treatment of trichotillomania has traditionally been Habit Reversal Training (HRT) (Twohig, Bluett, et al., 2014). Another form of treatment that is gaining empirical support is Acceptance and Commitment Therapy (ACT) which has been studied in four randomized controlled trials, one studying ACT as a standalone treatment (Lee, Homan, et al., 2018), and three examining ACT combined with HRT (Twohig et al., 2021; Lee, Haeger, et al., 2018; Woods, Wetterneck, et al., 2006) which demonstrated efficacy of the combined treatment in decreasing pulling symptom severity.

The prevalence of trichotillomania in the US is 1-2% of the population and yet treatment access is limited by many issues including processionals' lack of knowledge of the disorder and low treatment accessibility (Walther et al., 2010). ACT- enhanced behavior therapy has been implemented using telehealth to reach a larger population (42.2% decrease pre-to-post treatment), but telehealth still requires therapist time and incurs notable costs (Lee, Haeger, et al., 2018). The present study aims to address the gap in trichotillomania treatment accessibility by examining the role of check-ins on adherence and efficacy on afully automated, web-based ACT-enhanced HRT treatment for adults with trichotillomania across the United States. We predict that the condition with check-ins will increase adherence and efficacy of the treatment significantly more than the condition without check-ins. Additionally, we predict that hair pulling severity and psychological flexibility will be significantly improved by the condition with check-ins compared to the condition without check-ins.

ELIGIBILITY:
Inclusion Criteria:

1. Currently meet DSM-5 criteria for trichotillomania
2. searching for trichotillomania-based treatment
3. are atleast 18 years old
4. fluent English speakers
5. living in the U.S.

Exclusion Criteria:

1. currently receiving alternative therapy
2. currently modifying or starting psychotropic medication
3. previously met DSM-5 criteria for trichotillomania but are not, at the time of intake session, engaging in hair pulling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Massachusetts General Hospital- Hair Pulling Scale (MGH-HPS) | 36 weeks
  The MGH-HPS assesses urges to pull, pulling behavior, and the distress caused by pulling through a seven-item self-report measure. Items are rated individually on a scale from 0-4 and then the total scale is summed from 0-28-point total score. Higher scores indicate greater hair pulling severity. Treatment response is indicated by a seven-point reduction in score (Houghton et al., 2015). The MGH-HPS demonstrates good internal consistency (Keuthen et al., 1995), test-retest reliability and convergent and divergent validity (O'Sullivan et al., 1995).

CONTACTS AND LOCATIONS:
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided